CLINICAL TRIAL: NCT04048473
Title: : Assessment of Patient Satisfaction of Quality of Health Care Service and Treatment Provided by Outpatient Pain Management Clinic in Mansoura, Egypt.
Brief Title: Assessment of Patient Satisfaction of Quality of Health Care Service and Treatment
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, lecturer, Department of Anaesthesia, Intensive Care and pain management, Faculty of Medicine, Mansoura University
Other Study IDs: Assessment of Patient Satisfa
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MUH (Mansoura University Hospital): enrolled 127 patients in outpatient pain clinic The health service quality was assessed using Patient Satisfaction Questionnaire Short Form (PSQ-18) (ranging from strongly agree = 1, agree = 2, uncertain = 3, disagree = 4 and strongly disagree = 5). Also the treatment satisfaction using The Pain Treatment Satisfaction Scale (PTSS) was evaluated (ranging from 0 = dissatisfied to 100 = satisfied)
- Ocmu (Oncology center Mansoura University): enrolled132 patients in outpatient pain clinic The health service quality was assessed using Patient Satisfaction Questionnaire Short Form (PSQ-18) (ranging from strongly agree = 1, agree = 2, uncertain = 3, disagree = 4 and strongly disagree = 5).Also the treatment satisfaction using The Pain Treatment Satisfaction Scale (PTSS) was evaluated (ranging from 0 = dissatisfied to 100 = satisfied)

SUMMARY:
Patient satisfaction has become an important issue in the health services evaluation. It is equally important to medical results and economical costs of the provided services. Cancer is a common health problem frequently associated with pain that deserves patient satisfaction services. Assessment of patients' satisfaction in this sector of diseases is a cornerstone for optimum pain management. Recently, patient satisfaction is defined as personal evaluation of the experienced care, denoting both patient characteristics and care realities.

There are many questionnaires to assess patient satisfaction for health care service and treatment. For health service assessment, Patient Satisfaction Questionnaire Short Form (PSQ-18) is a commonly used one with high reliability. It includes seven dimensions of patient satisfaction which are general satisfaction, interpersonal manner, communication, technical quality, time spent with doctor, financial aspects, and accessibility and convenience.

With regard to patient satisfaction about the provided treatment, Pain Treatment Satisfaction Scale (PTSS) is routinely applied.

It is well known that any health care system needs continuous evaluation both by the care givers and patients in order to improve the quality of service. Of course, it is a continuous process with much variability. There are many studies about patient satisfaction in cancer patients., however this study is the first in Delta region, Egypt. From this point, the aim of this study is to evaluate the quality offered by health care services and the treatment satisfaction among cancer patients attending the outpatient pain management clinics, Mansoura, Egypt in two university centers.

DETAILED DESCRIPTION:
It is a cross sectional comparative study in the outpatient pain clinic of MUH and OCMU. These centers serve Delta Region which encompasses 10 governorates with 41% of the total Egyptian population. The study was approved by the Institutional Research Board (Code No: R.19.04.480 ). The sample was recruited using convenience sampling method during the period from April 2019 till July 2019. Two hundred fifty nine patients received medical care with chronic cancer pain aged 18 years or older that are oriented, alert, speak and read Arabic, having no communication problems or physical conditions that will prevent the completion of the interview were included in this study. Patients do not speak or read Arabic, or who are unable to complete the study questionnaires were excluded.

Physicians screen patients for suitability in the study and consent those who met the inclusion criteria. During the studies, participants complete the paper of the measures while they are waiting for their medical consultation.

The health service quality was assessed using Patient Satisfaction Questionnaire Short Form (PSQ-18) (ranging from strongly agree = 1, agree = 2, uncertain = 3, disagree = 4 and strongly disagree = 5). It contains seven domains; general satisfaction (questions (Q) 3 &17), technical quality(Q 2,4,6 &14), interpersonal manner (Q 10& 11), communication (Q 1 & 13), financial aspects (Q 5&7), time spent with the doctor (Q12&15) and accessibility and convenience (Q 8,9,16 &18).4 Also we evaluated the treatment satisfaction using The Pain Treatment Satisfaction Scale (PTSS) (ranging from 0 = dissatisfied to 100 = satisfied): It includes thirty nine items grouped into five dimensions; satisfaction with current pain medication in two subscales: medication characteristics (3 items) and efficacy (3 items); side effects of medication (12 items); impact of current pain medication (8 items); medical care (8 items) and information about pain and its treatment (5 items).

ELIGIBILITY:
Inclusion Criteria:

* patients received medical care with chronic cancer pain
* aged 18 years or older
* oriented, alert,
* speak
* read Arabic,
* having no communication problems
* having nophysical conditions that will prevent the completion of the interview

Exclusion Criteria:

* Patients do not speak
* Patients do notread Arabic,
* are unable to complete the study questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred fifty nine patients received medical care with chronic cancer pain aged 18 years or older that are oriented, alert, speak and read Arabic, having no communication problems or physical conditions that will prevent the completion of the interview were included in this study.
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
The Pain Treatment Satisfaction Scale (PTSS) | during the 1 day visit
  (ranging from 0 = dissatisfied to 100 = satisfied)It includes thirty nine items grouped into five dimensions; satisfaction with current pain medication in two subscales: medication characteristics (3 items) and efficacy (3 items); side effects of medication (12 items); impact of current pain medication (8 items); medical care (8 items) and information about pain and its treatment (5 items).
Patient Satisfaction Questionnaire Short Form (PSQ-18). | during the 1 day visit
  (ranging from strongly agree = 1, agree = 2, uncertain = 3, disagree = 4 and strongly disagree = 5). It contains seven domains; general satisfaction (questions (Q) 3 &17), technical quality(Q 2,4,6 &14), interpersonal manner (Q 10& 11), communication (Q 1 & 13), financial aspects (Q 5&7), time spent with the doctor (Q12&15) and accessibility and convenience (Q 8,9,16 &18)

SECONDARY OUTCOMES:
Pain intensity in the present, average and the worst pain using Numerical Rating Scale (NRS) | during the 1 day visit
  It is an 11-point scale that 0 (no pain) and 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Nevert Adel Abdel Ghaffar, Al Mansurah, Egypt